CLINICAL TRIAL: NCT06561399
Title: A Single-arm, Phase II, Prospective Study of Transcatheter Arterial Chemoembolization, Lenvatinib Combination With Sintilimab Sequential Radiotherapy in Patients With Initial Unresectable Hepatocellular Carcinoma
Brief Title: Triple Therapy Sequential Radiotherapy in Unresectable HCC (TALENP003)
Status: Recruiting | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ming Wei, Department of Hepatobiliary Pancreatic Surgery, Fujian Provincial Hospital
Other Study IDs: TALENP003
Record Dates: First submitted 2024-07-13; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular carcinoma; TACE; Lenvatinib; Sintilimab; radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Triple Therapy sequential Radiotherapy
  Interventions: Combination Product: TACE, Lenvatinib combination with Sintilimab sequential radiotherapy

INTERVENTIONS:
Combination Product: TACE, Lenvatinib combination with Sintilimab sequential radiotherapy — TACE, Lenvatinib [8mg(<60kg)/12mg(>60kg) orally daily] combination with Sintilimab (200mg administered intravenous injection on Day 1 of each 21-day cycle) for 2 months. Sequential radiotherapy method and dosage are comprehensively evaluated by radiologists, hepatobiliary surgeons, and oncologists, and discussed by a multidisciplinary team

SUMMARY:
This is an Open-label, Multicenter, Phase II clinical trial to evaluate the efficacy and safety of Transcatheter arterial chemoembolization (TACE), Lenvatinib combination with Sintilimab (Triple Therapy) sequential radiotherapy in patients with Unresectable Hepatocellular Carcinoma (uHCC).

DETAILED DESCRIPTION:
For Unresectable Hepatocellular Carcinoma (uHCC) patients, Transcatheter arterial chemoembolization (TACE), Lenvatinib combined with PD-1 inhibitors treatment is an important choice, which can achieve deeper tumor remission. However, there are still some patients whose lesions have not reached complete response after treatment. According to research, patients with complete response of lesions after conversion therapy have a more ideal long-term survival rate. For populations that have not yet achieved complete response, sequential radiotherapy will achieve deeper tumor remission, delay recurrence, and achieve better oncological outcomes. This study is a single arm, multicenter, prospective clinical trial designed to evaluate the efficacy and safety of TACE, Lenvatinib combination with Sintilimab (Triple Therapy) sequential radiotherapy in the treatment of uHCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to enrollment in this study, signing the informed consent form;
2. Age between 18 and 75 years old, male or female patients;
3. Child-Pugh class A;
4. Indocyanine green 15 min retention rate (ICGR-15) <15%;
5. ECOG score 0-1;
6. Diagnosis of hepatocellular carcinoma according to the Chinese HCC Diagnosis and Treatment Guidelines 2022 Edition and expected survival time greater than 4 months.
7. Patients with a diagnosis of initial unresectable HCC (BCLC stage B or C), evaluated as partial response (PR) or stable disease (SD) by RECIST 1.1 after 2 months of treatment with TACE, Lenvatinib combination with Sintilimab. The number of residual active lesions in the liver was 1 to 3 and suitable for radiation therapy. Fusion lesions in the liver were considered as 1 lesion, and portal vein cancer thrombus was considered as 1 lesion for treatment.
8. Normal tissue limits were performed according to the UK Consensus on Normal Tissue Dose Constraints for Stereotactic Radiotherapy.
9. Patients who have not received any tumor-related targeted, immunotherapy, radiotherapy and chemotherapy before enrollment;
10. Patients with at least one measurable lesion according to RECIST 1.1 criteria (measurable lesion CT/MRI scan length diameter ≥10mm, and measurable lesion has not received localized treatments such as radiotherapy, cryotherapy, etc.);
11. Blood routine: absolute neutrophil count ≥1.5×10^9/L, Hb ≥8.5g/L, PLT ≥75×10^9/L;
12. No history of severe cardiac arrhythmia or heart failure; no history of severe ventilatory dysfunction or severe pulmonary infection; no acute or chronic renal failure with creatinine clearance >40 mL/min;
13. Women of childbearing age should agree that they must use contraception during and for 6 months after the end of the dosing period; patients who have had a negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating, and men should agree that they must use contraception during and for 6 months after the end of the study period.

Exclusion Criteria:

1. Patients with a diagnosis of initial unresectable HCC, assessed as complete response (CR) or Progressive disease (PD) by RECIST 1.1 after 2 months of treatment with TACE, Lenvatinib combined with Sintilimab;
2. Tumor combined with cancerous thrombus in the inferior vena cava and the tumor has developed extrahepatic metastasis;
3. Treatment with other antitumor therapy such as targeted drugs, PD-1/PD-L1 inhibitors, surgery, TACE, radiotherapy, FOLFOX systemic chemotherapy, and locus coeruleus granule drugs prior to study entry;
4. History of allergy to Lenvatinib, Sintilimab and their components;
5. Tumor volume accounting for two-thirds or more of the liver volume or diffuse distribution of intrahepatic lesions;
6. Presence of any active autoimmune disease or patients with autoimmune disease with expected relapse (e.g., interstitial pneumonitis, colitis, hepatitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including, but not limited to, these disorders and syndromes); hypothyroidism treated with stabilized doses of thyroid-replacing hormone; 1-year old diabetes mellitus using stabilized doses of insulin; or Type 1 diabetes mellitus; but not vitiligo or resolved childhood asthma/allergies that do not require any intervention in adulthood;
7. Patients have history of immunodeficiency; patients who are on immunosuppressive or systemic hormone therapy for immunosuppression and have continued to do so within 2 weeks prior to signing the informed consent form
8. Have known hereditary or acquired bleeding (e.g., coagulation disorders) or thrombotic tendencies, such as in patients with hemophilia; current or recent (within 10 days prior to initiation of study treatment) use of full-dose oral or injectable anticoagulant or thrombolytic medications for therapeutic purposes (prophylactic use of low-dose aspirin, low-molecular heparin is permitted)
9. Severe infections (CTCAE > Grade 2) such as severe pneumonia requiring hospitalization, bacteremia, or infectious co-morbidities within 4 weeks prior to the first dose of study drug; baseline chest imaging suggestive of active lung inflammation, signs and symptoms of infection within 2 weeks prior to the first dose of study drug, or requiring treatment with oral or intravenous antibiotics (excluding prophylactic antibiotics). (excluding prophylactic use of antibiotics);
10. Patients with proteinuria with routine urinalysis suggestive of ≥ 1 + will undergo a 24-hour urine protein test for 24-hour urine protein ≥ 1g;
11. Have history of other malignant tumors within the previous 5 years or concurrently, except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix and papillary thyroid carcinoma;
12. Patients with co-morbid mental diseases; history of psychotropic substance abuse, alcoholism and drug addiction;
13. Women who are pregnant or breastfeeding
14. Patients with obvious contraindications to surgery, such as renal and cardiopulmonary insufficiency, as judged by the investigator, and those who, in the opinion of the investigator, should not participate in this trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Unresectable Hepatocellular Carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | 4 weeks after the initiation of medication until the day before surgery
  The objective response rate (ORR) was defined as the complete response (CR) rate + the partial response (PR) rate according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression free survival, PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The Progression free survival (PFS) was defined as the time between the start of treatment and the progression of intrahepatic and/or extrahepatic tumors, or the occurrence of death or loss of follow-up for any reason.
Overall survival, OS | From date of randomization until the date of death from any cause, whichever came first, assessed up to 60 months
  The Overall survival (OS) was defined as the time between receiving treatment and observing death or loss of follow-up for any reason.
Objective response rate, ORR | 4 weeks after the initiation of medication until the day before surgery
  The objective response rate (ORR) was defined as the complete response (CR) rate + the partial response (PR) rate according to mRECIST.
Conversion resection rate, CRR | 3 months
  The Conversion resection rate (CRR) was defined as the patient who reach the resectable criterion after treatment and accepted operation.
Major pathological response rate, MPR rate | Immediately after surgery
  The major pathological response (MPR) rate was defined as less than 10% active tumor cells in the excised tissue sample in patients accept operation.
Toxicity Adverse events | through study completion, assessed up to 60 months
  Grade 1-5 AEs according to NCI-CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Ming Wei, Principal Investigator — Fujian Provincial Hospital
Locations (4):
- China (4):
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Fujian provincial hospital, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian

IPD SHARING:
Plan to Share IPD: No